CLINICAL TRIAL: NCT07041593
Title: The Effect of Inspiratory Muscle Training on Functional Gain in Cerebral Palsy: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sadık Emre ÇELEBİ (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Medipol University (Other)
Responsible Party: Sponsor-Investigator, Sadık Emre ÇELEBİ, MSc, PhD(c), Physiotherapist, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-202.3.02-2938
Record Dates: First submitted 2025-06-16; First posted 2025-06-27 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy; Respiratory Muscle Training; Dysphagia; Balance Control; Functional Abilities; Respiratory Function Test
Keywords: Cerebral Palsy; Respiratory muscle training; Inspiratory muscle traning; Trunk control; Swallowing disorder; Upper extremity functionality
MeSH Terms: conditions — Cerebral Palsy; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will undergo a traditional physiotherapy programme for 8 weeks, consisting of two 40-minute sessions per week under the supervision of a physiotherapist.
  Interventions: Other: Traditional Physiotherapy
- Experimental Group (Experimental): Participants in this group will receive inspiratory muscle training (IMT). IMT will be performed twice a week under the supervision of a physiotherapist and as a home exercise programme on the remaining days, for a total of eight weeks, five days a week, for 15 minutes a day. In addition, participants will receive traditional physical therapy treatments. In addition, participants will undergo an 8-week traditional physiotherapy programme consisting of two 40-minute sessions per week under the supervision of a physiotherapist.
  Interventions: Other: Inspiratory Muscle Training and Traditional Physiotherapy

INTERVENTIONS:
Other: Inspiratory Muscle Training and Traditional Physiotherapy — Participants in this group will undergo inspiratory muscle training (IMT). The resistance to be applied at the start of IMT has been set at 30% of the maximum inspiratory pressure (MIP) value. The MIP value will be remeasured every week, and the training load will be updated according to 30% of the new value obtained. IMT will be carried out twice a week with a physiotherapist and on the remaining days as a home programme, for a total of eight weeks, five days a week, 15 minutes a day. Participants in the experimental group will receive traditional physical therapy treatments for cerebral palsy in the same manner as the control group. In this context, traditional physical therapy methods based on neurodevelopmental principles will be applied and designed according to the individual's needs.
  Arms: Experimental Group
Other: Traditional Physiotherapy — Participants in the control group will undergo a neurodevelopmental-based traditional physiotherapy programme for 8 weeks, with two 40-minute sessions per week under the supervision of a physiotherapist; on other days, they will be asked to continue the exercises taught to their families at home.
  Arms: Control Group

SUMMARY:
This study investigates the effect of respiratory muscle training on respiratory muscle strength, respiratory parameters, trunk control, upper extremity function and dysphagia in patients with cerebral palsy aged 5-18 years. The results of the study aim to provide a clinical perspective for clinicians working with patients diagnosed with cerebral palsy between the ages of 5-18 years and to contribute to the literature.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a neurodevelopmental disorder characterised by permanent motor dysfunctions that develop in the prenatal, perinatal or postnatal period as a result of nonprogressive central nervous system involvement. CP involves not only the musculoskeletal system but also many different systems such as respiratory, digestive, sensory and cognitive systems, leading to a complex involvement. The complex involvement associated with the nature of CP necessitates a holistic and multidisciplinary approach in terms of treatment. In addition to common motor dysfunctions in the clinical picture, common comorbidities include epilepsy, swallowing disorders (dysphagia), gastrointestinal problems (e.g. constipation and reflux), nutritional deficiencies, behavioural problems, sensory disorders and respiratory system complications.

In individuals with CP, musculoskeletal system involvement results in significant comorbidities in the respiratory system. Especially weakness of respiratory muscles, inadequate airway clearance, increased risk of aspiration and recurrent respiratory tract infections are among the important complications reported in individuals with CP. This situation is more prominent especially for patients at levels IV and V according to the Gross Motor Function Classification System (GMFCS) and significantly negatively affects the quality of life of both the individual with CP and their caregivers.

Another important dysfunction in patients with CP is dysphagia, which develops mostly due to impaired motor control and coordination in the oral and pharyngeal phases. Oropharyngeal dysphagia (OPD) is quite common in children with CP and may lead to serious complications such as aspiration, malnutrition, growth retardation, gastroesophageal reflux disease and pneumonia. This effect, which can be seen in all phases of swallowing disorders, causes a decrease in muscle mass and immune functions by reducing energy intake, which increases susceptibility to infection.

In the field of pulmonary rehabilitation, individualised exercise programmes targeting respiratory muscles have recently attracted considerable attention, and studies using inspiratory muscle training (IMT) and feedback devices have provided significant improvements in maximum inspiratory and expiratory pressures. Studies have reported significant increases in daily living activities and quality of life of individuals after respiratory muscle training.

In line with the literature, the aim of this study was to investigate the effect of respiratory muscle training on respiratory muscle strength, respiratory and swallowing functions of individuals diagnosed with CP. In addition to the parameters mentioned in the study, the effectiveness of respiratory muscle training on trunk control and upper extremity functions in individuals with CP will also be questioned.

ELIGIBILITY:
Inclusion Criteria:

* Level I or II according to the Gross Motor Function Classification System (GMFCS)
* Communication skills sufficient to understand spoken or written language
* Diagnosed with cerebral palsy (CP) by a paediatric neurologist
* Aged between 5 and 18 years old
* Participants whose families have given written consent to participate in the study will be included in the study.

Exclusion Criteria:

* Those who have had a respiratory tract infection within the last month,
* Those with haemodynamic instability (heart rate > 150 beats/minute, systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg),
* Those who have undergone orthopaedic surgery or botulinum toxin injection within the last six months,
* Participants with severe chest infections or existing respiratory problems that would prevent them from participating in the study,
* Participants with mental or auditory dysfunction that would prevent them from participating in the assessment and intervention processes are planned to be excluded from the study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory pressure assessment | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  For the measurement of maximum inspiratory pressure (MIP), participants will be asked to first exhale against a valve that closes the airway, and then perform maximum inspiration. Measurements will be terminated when the difference between three consecutive trials is less than 10 cmH₂O. The highest MIP value will be selected for use in analyses.

SECONDARY OUTCOMES:
Maximum expiratory pressure assessment | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  In the maximum expiratory pressure (MEP) measurement, subjects will first inhale and then exhale as hard as they can against the valve. Measurements will be terminated when the difference between three consecutive trials is less than 10 cmH₂O. The highest MEP value will be selected for use in the analyses.
Assessment of upper extremity function | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  The AbilHand-Kids questionnaire will be used to assess participants' upper extremity function in daily life. The questionnaire is a 21-item survey that evaluates children's upper extremities bilaterally and assesses their ability to perform common tasks in daily living activities. The maximum score that can be obtained from the questionnaire is 42, and the minimum score is 0. A high score indicates that the individual uses their hand better in daily life compared to those with lower scores. An increase in the score indicates positive development, while a decrease in the score indicates negative development.
Assessment of swallowing | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  The Pediatric Eating Assessment Tool-10 (PEDI-EAT-10) will be used to assess dysphagia. This 10-item scale is scored on a scale of 0-4 for each item. High scores on the scale are considered to indicate a risk of swallowing disorder or severe dysphagia symptoms.
Assessment of trunk control | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  The Trunk Control Measurement Scale will be used to assess participants' trunk control. This scale assesses trunk control during functional activities. The scale contains a total of 15 items. The total score on the scale ranges from 0 to 58 points, with higher scores indicating better performance.
Forced vital capacity (FVC) massessment | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be recorded in litres.
Forced expiratory volume in one second (FEV1) assessment | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be recorded in litres.
FEV1/FVC ratio | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  FVC and FEV1 results will be compared and expressed as percentages.
Forced expiratory flow 25-75% (FEF25-75) assessment | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be expressed in litres per second.
Peak expiratory flow (PEF) assessment | The first assessment will be conducted during the first week. The final assessment will be conducted after the 8-week intervention.
  Patients will perform a rapid and complete inhalation maneuver from functional residual capacity to total lung capacity, followed by a continuous and maximal exhalation maneuver lasting at least six seconds. Verbal and non-verbal encouragement will be provided throughout the maneuvers. The test will be terminated once acceptable repeatability is achieved. The results will be expressed in litres per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Sadık E Çelebi, MSc, PhD(c), Physiotherapist, Study Chair — Istanbul University-Cerrahpaşa, Cardiology Institute, Department of Cardiology
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol